CLINICAL TRIAL: NCT00290810
Title: A Phase II Trial of Bevacizumab to Prevent or Delay Disease Progression in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: Bevacizumab in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00137; NCI-2009-00137 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MC048C; NCI-7211; CDR0000459933; MC048C (Other: Mayo Clinic); 7211 (Other: CTEP); P30CA015083 (NIH); N01CM62205 (NIH); N01CM62207 (NIH); NCT01646996 (obsolete NCT alias); NCT01664364 (obsolete NCT alias)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2013-05-14 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2012-04

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bevacizumab

ARMS (1):
- Treatment (monoclonal antibody therapy) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
This phase II trial is studying how well bevacizumab works in treating patients with relapsed or refractory B-cell chronic lymphocytic leukemia. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bevacizumab may also stop the growth of cancer cells by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the treatment success rate of Bevacizumab in patients with relapsed or refractory B-cell chronic lymphocytic leukemia (CLL).

II. Assess the toxicity associated with this regimen in patients with relapsed or refractory CLL

SECONDARY OBJECTIVES:

I. Assess sensitivity to apoptosis/cell death of residual B-cell clone during therapy (e.g. is treatment selecting out a resistant clone).

II. Evaluate if the risk stratification parameters (ie immunoglobulin mutational, ZAP-70, FISH defects and /or CD38 status) corresponds to both baseline apoptosis/cell death and the rates of apoptosis of CLL B-cells when cultured with Bevacizumab.

III. Examine if Bevacizumab can be synergistic with other chemotherapeutic drugs such as chlorambucil or fludarabine.

IV. Assess if marrow vascularity is increased at entry to study and if it is modulated following therapy with Bevacizumab.

V. Examine the association of VEGF plasma levels at baseline with clinical responses to Bevacizumab.

VI. Examine the levels of VCAM at entry to the study and during treatment with Bevacizumab.

OUTLINE: This is a multicenter study. Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15.

Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL)*, as defined by the following phenotypic characteristics:

  * Predominant population of cells share both B-cell antigens (CD19, CD20, or CD23) as well as the T-cell antigen (CD-5), in the absence of other pan-T-cell markers (CD-3, CD-2, etc.)

    * Mantle cell lymphoma must be excluded by demonstrating the absence of the t(11;14) by fluorescent in situ hybridization (FISH)
  * Dim surface immunoglobulin expression
  * Exclusively kappa and lambda light chains
* Peripheral blood absolute lymphocyte count > 5,000/mm^3

  * Lymphocytosis must consist of small to moderate size lymphocytes, with ≤ 55% prolymphocytes, atypical lymphocytes, or lymphoblasts morphologically
* Requires chemotherapy, as indicated by any of the following:

  * Disease related symptoms, including the following:

    * Weight loss ≥ 10% within the previous 6 months
    * Extreme fatigue
    * Fevers > 100.5°F for 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Evidence of progressive marrow failure, as manifested by the development of or worsening anemia (hemoglobin ≤ 10 g/dL) and/or thrombocytopenia (platelet count ≤ 100,000/mm^3)
  * Massive (i.e., > 6 cm below left costal margin) or progressive splenomegaly
  * Measurable and progressive lymphadenopathy
  * Measurable (i.e., > 5,000/mm^3) and progressive lymphocytosis
* Progressive disease or relapsed after or refractory to 1 course of an alkylating agent-based or purine nucleoside-based (e.g., fludarabine) regimen
* No marrow function attributable to dysplasia related to prior therapy
* ECOG performance status 0, 1, or 2
* Serum creatinine < 2 mg/dL

  * If serum creatinine > 1.5 mg/dL but < 2 mg/dL, creatinine clearance must be ≥ 30 mL/min
* Platelet count > 30,000/mm^3
* Direct bilirubin ≤ 2 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other second malignancy within the past 2 years except squamous cell or basal cell carcinoma of the skin or in situ carcinoma of the cervix
* No New York Heart Association class III or IV heart failure
* No blood pressure > 150/90 mm Hg
* No unstable angina
* No myocardial infarction or stroke within the past 6 months
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 28 days
* Urine protein:creatinine (UPC) ratio ≤ 1.0

  * Patients with a UPC ratio > 1.0 must undergo a 23-hour urine collection and must demonstrate < 1 gram of protein per day
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious, non-healing wound, ulcer, or bone fracture
* No active infections requiring oral or intravenous antibiotics
* No active bleeding or pathological conditions that carry a high risk of bleeding (e.g., known varices)
* No thrombocytopenia requiring transfusion
* See Disease Characteristics
* More than 4 weeks since prior participation in an experimental drug study
* At least 8 weeks since prior rituximab
* At least 6 weeks since prior chemotherapy
* More than 28 days since prior major surgery or open biopsy
* More than 7 days since prior minor surgery, fine needle aspirations, or core biopsies
* No concurrent major surgery
* No concurrent participation in another experimental drug study
* Concurrent full-dose warfarin or low molecular weight heparin allowed provided patient is on a stable dose AND INR is in range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-12; Primary Completion 2008-10 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tait Shanafelt, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen patients were accrued to the bevacizumab trial between December 2005 and March 2009.
Pre-assignment Details: One patient never received protocol treatment due to a high protein:creatinine ratio and high 24-hour urine protein excretion. Accordingly, 12 eligible patients were included in the outcome analysis.
Period: Overall Study
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 73 [60 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Confirmed Objective Status of Complete Response (CR), Complete Clinical Response (CCR), Nodular Partial Response (nPR), or Partial Response (PR).
Description: The NCI Working Group criteria will be used to assess response to therapy. A confirmed response is defined as a response documented on 2 consecutive evaluations at least 4 weeks apart.
  Complete Response:
  * No lymphadenopathy
  * No hepatomegaly or splenomegaly
  * Absense of constitutional symptoms
  * Polymorphonuclear leukocytes ≥ 1500/ul
  * Platelets > 100,000/ul
  * Hemoglobin > 11.0 gm/dl
  * Peripheral blood lymphocytes ≤ 4000/uL.
  * Confirmation by Marrow Aspirate and biopsy.
  Complete Clinical Response:
  -CR without bone marrow biopsy confirmation.
  Nodular Partial Response:
  -CR with the presence of residual clonal nodules.
  Partial Response requires:
  * ≥ 50% decrease in peripheral blood lymphocyte count
  * ≥ 50% reduction in lymphadenopathy
  * ≥ 50% reduction in size of liver and/or spleen
  * 1 or more of the following:
    * Polymorphonuclear leukocytes ≥ 1500/ul
    * Platelets >100,000/ul
    * Hemoglobin >11.0 gm/dl
Time Frame: Up to 5 years
Population: All 12 patients are used in this analysis
Measure: Number; unit: participants
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 12
participants
  Complete Response (CR) | 0
  Complete Clinical Response (CCR) | 0
  Nodular Partial Response (nPR) | 0
  Partial Response (PR) | 0

2. Secondary Outcome: Toxicity Associated With This Regimen in Participants With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL).
Description: As per NCI Common Toxicity Criteria for Adverse Effects (CTCAE) Version 3.0, the term toxicity is defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment. The number of participants experiencing grade 3 or higher toxicity will be reported here.
Time Frame: From the date of registration to the to the date of last treatment evaluation, median number of days on treatment was 56 days.
Population: All 12 participants treated will be used to analyze this endpoint.
Measure: Number; unit: participants
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 12
participants
  Grade 3 Toxicity | 5
  Grade 4 Toxicity | 1

3. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method will be used to estimate distributions in the B-CLL population.
Time Frame: From the date of registration to the date of the event (i.e., death or the date of last follow-up), up to 5 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 12
months | 39.75 [5.65 to NA] — Too few events occurred to obtain an estimate.

4. Secondary Outcome: Time to Progression
Description: Progression is defined as one of the following:
  * A ≥50% increase in the sum of the products of at least 2 lymph nodes on 2 consecutive determinations 2 weeks apart (at least one node must be ≥2 cm) or the appearance of new palpable lymph nodes, or
  * A ≥50% increase in the size of the liver and/or spleen as determined by measurement below the respective costal margin or the appearance of hepatomegaly or splenomegaly which was not previously present, or
  * The transformation to a more aggressive histology (e.g. Richter's transformation), or
  * A ≥ 50% increase in the absolute number of circulating lymphocytes.
  The Kaplan-Meier method will be used to estimate time to progression.
Time Frame: From the date of registration to the date of the event (i.e., death or disease progression) or the date of last follow-up, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 12
months | 2.9 [1.8 to 3.7]

ADVERSE EVENTS:
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody Therapy) (N=12)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Eye disorder (Eye disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody Therapy) (N=12)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (5)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (12)
Fever (General disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 4 (5)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (3)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (6)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less